CLINICAL TRIAL: NCT03649126
Title: Nationwide Implementation of Standardized Structured Reporting to Support Optimal Treatment Decisions
Brief Title: Nationwide Implementation of Standardized Structured Reporting
Acronym: IMPROVING
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other); PALGA foundation (Other)
Responsible Party: Principal Investigator, Rosella Hermens, dr., Radboud University Medical Center
Other Study IDs: KWF-8281; 2018-4124 (Other: CMO - Radboudumc)
Record Dates: First submitted 2018-08-14; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Standardized Structured Reporting
Keywords: standardized structured reporting; treatment decisions; multidisciplinary team; pathology; implementation tools

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Dutch pathologists hospital I: Pathologists in hospital I using protocols of:
  Urological cancer Gynaecological cancer Gastro intestinal cancer
  Interventions: Behavioral: Implementation tools
- Dutch pathologists hospital II: Pathologists in hospital II using protocols of:
  Urological cancer Gynaecological cancer Gastro intestinal cancer
  Interventions: Behavioral: Implementation tools
- Dutch pathologists hospital III: Pathologists in hospital III using protocols of:
  Urological cancer Gynaecological cancer Gastro intestinal cancer
  Interventions: Behavioral: Implementation tools
- Dutch pathologists hospital IV: Pathologists in hospital IV using protocols of:
  Urological cancer Gynaecological cancer Gastro intestinal cancer
  Interventions: Behavioral: Implementation tools
- Dutch pathologists hospital V: Pathologists in hospital V using protocols of:
  Urological cancer Gynaecological cancer Gastro intestinal cancer
  Interventions: Behavioral: Implementation tools
- Dutch pathologists hospital VI: Pathologists in hospital VI using protocols of:
  Urological cancer Gynaecological cancer Gastro intestinal cancer
  Interventions: Behavioral: Implementation tools

INTERVENTIONS:
Behavioral: Implementation tools — Implementation tools developed by experts in order to increase the use of SSR in pathology

SUMMARY:
The first objective is to explore factors that impede or facilitate implementation of SSR in pathology (and other disciplines) among the MDT members receiving SSRs. The second objective is to select, develop and evaluate (process and effect outcomes) implementation tools supporting optimal implementation of SSR in pathology. The third objective is to offer implementation tools to all pathology laboratories in the Netherlands and to share the SSR-kit for successful implementation with other medical disciplines

DETAILED DESCRIPTION:
By implementing SSR in various disciplines, we contribute to improving communication, efficiency and quality of multidisciplinary team (MDT) meetings and facilitate optimal treatment decision making. Optimal discussion of each patient at MDT meetings can be achieved by a clear communication of all diagnostic results among MDT members. However, the adoption of innovations, such as SSR, is laborious, especially when the innovation requires changing daily habits. Offering implementation tools supports the adoption of innovations among medical professionals. Implementation tools are most effective when they are developed on the basis of factors that impede or facilitate the innovation. Besides the importance of investigating these factors for SSR among pathologists, we will also involve MDT members receiving pathology SSRs in our study. After all, because MDT members will greatly benefit from SSR, they could play a key role in stimulating the use of SSR among pathologists. Therefore, we will also explore which tools MDT members need to stimulate the diagnostic disciplines in using SSR. Subsequently, we will develop and evaluate implementation tools to support the use of SSR by pathologists. The kit for successful implementation of SSR will be offered to other medical disciplines like radiology, endoscopy, and surgery who face similar challenges with implementation of SSR. The SSR-kit consists of our multidisciplinary approach for the whole process of developing implementation tools for SSR, examples of tools for SSR, and other results of this project.

ELIGIBILITY:
Inclusion Criteria:

* Pathologists of urological, gynecological or gastro-intestinal cancers
* Other MDT-members of urological, gynecological or gastro-intestinal cancers (medical oncologists, radiologists, radiotherapists, urologists, gynecologists, intestinal surgeons, nuclear medicine physicians, nurse practitioners).
* Dutch
* Residents

Exclusion Criteria:

* Retirees

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dutch pathologists, MDT-members and residents, using SSR of urological, gynecological or gastro-intestinal cancers.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-21 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Barriers and facilitators in implementation of SSR in MDT - focus groups and self-developed questionnaire | 9 months
  Barriers and facilitators in implementation of SSR among MDT members measured by focus groups and a self-developed questionnaire
Effectiveness of implementation tools - frequencies of use of SSR templates in pathology in the Netherlands | 6 months
  The improvement in use of SSR templates in the Netherlands (=effectiveness of implementation tools) measured by frequencies of use of SSR templates in pathology (=all laboratories in the Netherlands)

SECONDARY OUTCOMES:
Determinants of barriers and facilitators in implementation of SSR - focus groups and a self-developed questionnaire | 1 month
  Determinants of barriers and facilitators in implementation of SSR among MDT members measured by focus groups and a self-developed questionnaire
Experiences with implementation tools - questionnaire | 6 months
  Experiences of pathologists and other MDT members with the implementation tools, measured by a questionnaire
Use of implementation tools - questionnaire | 6 months
  Use of implementation tools among pathologists and other MDT members, measured by a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided